CLINICAL TRIAL: NCT00152867
Title: A Randomised Double-Blind Placebo Controlled Cross Over Trial of the Impact on Quality of Life of Continuing Dexamethasone Beyond 24 Hours Following Moderately Emetogenic Chemotherapy
Brief Title: Dexamethasone Study: Impact on Quality of Life of Continuing Dexamethasone Following Emetogenic Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Ian Tannock, University Health Network
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MDJV2
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Cancer; Emesis; Nausea
Keywords: quality of life; dexamethasone; emesis
MeSH Terms: conditions — Neoplasms; Vomiting; Nausea | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Dexamethasone
  Interventions: Drug: Dexamethasone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — dexamethasone 4mg PO bd for 2 days post chemotherapy

SUMMARY:
Background: Dexamethasone is a steroid, which is often given into the vein before chemotherapy to help control acute nausea and vomiting. It can also be given as an oral tablet for patients to take for the two days following chemotherapy to help minimise delayed nausea and vomiting. In chemotherapy regimens that cause high rates of nausea and vomiting, the use of dexamethasone is well proven. However, in chemotherapy regimens that generally cause only minimal to moderate rates of nausea and vomiting, the value of oral dexamethasone in the 48-hour period after chemotherapy is not well proven, although it is often prescribed. While dexamethasone does decrease nausea, it causes additional side-effects such as insomnia, indigestion, anxiety and mood changes. While patients with less vomiting and nausea are expected to have better quality of life (QOL), for patients with minimal nausea or vomiting, their QOL might be more affected by the side effects of the dexamethasone treatment than by the nausea.

Study Design: The study will be performed in patients who will be receiving first line chemotherapy treatment with a moderate risk of nausea/vomiting. Anti-nausea therapy for acute nausea/vomiting will be standardised and all patients will receive non-steroidal medication for delayed nausea control. Each patient will be randomly allocated to receive either oral dexamethasone or an identical appearing placebo tablet for two days after chemotherapy for the first cycle of chemotherapy, and then crossed over to the other treatment for the second cycle. Patients will complete QOL assessments, dexamethasone symptom and nausea and vomiting questionnaires, as well as nausea/vomiting diaries. This will enable the researchers to determine the effect of dexamethasone on nausea and vomiting and the impact of both the side effects of dexamethasone, and of nausea and vomiting, on QOL.

Objectives: The primary objectives are to determine patient preference for dexamethasone or placebo, and to compare changes in QOL after chemotherapy in patients who receive dexamethasone with those who receive placebo. The secondary objectives are: (1) to compare complete protection from delayed vomiting and severity of nausea; (2) to compare differences in the impact of nausea and vomiting on QOL, and (3) to compare differences in symptoms that have been associated with dexamethasone (insomnia, anxiety, agitation, mood, etc.) between patients receiving dexamethasone and those receiving placebo.

Significance: This study will provide data to evaluate whether the benefits of dexamethasone for delayed nausea and vomiting outweigh potential side effects in patients receiving chemotherapy with a moderate risk of causing nausea and vomiting. This addresses a problem that is important to a majority of patients receiving anticancer chemotherapy. If overall QOL is improved on dexamethasone, then it should be prescribed more frequently, but if QOL is reduced on dexamethasone, and patients prefer the placebo, then its use as an anti-nausea medication for delayed nausea after moderately nauseating chemotherapy should be limited to patients with poor initial control of nausea/vomiting.

DETAILED DESCRIPTION:
Background: Dexamethasone improves control of acute nausea and vomiting when given prior to chemotherapy, and continued administration of dexamethasone improves nausea and vomiting after highly emetogenic chemotherapy. There is no consensus about the optimal regimen for control of delayed emesis after moderately emetogenic chemotherapy but most patients receive oral dexamethasone. Many patients complain of insomnia, anxiety/agitation and indigestion whilst they are on dexamethasone, and fatigue and depressed mood after stopping it. The impact of these symptoms on patients has not been studied systematically. While patients with less vomiting and nausea are expected to have better quality of life (QOL), the QOL of patients with minimal nausea or vomiting might be more affected by the side effects of antiemetic treatment.

Hypothesis: Dexamethasone given as an antiemetic for delayed nausea and vomiting after moderately emetogenic chemotherapy reduces overall quality of life.

Research Question: Does the use of dexamethasone as a prophylactic antiemetic for delayed nausea and vomiting following moderately emetogenic chemotherapy decrease overall quality of life, as evaluated by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C-30).

Study Design: Using a double-blind randomised cross-over design, we will determine:

* (i) the effect of oral dexamethasone (4mg PO bid after chemotherapy) versus an identical appearing placebo on QOL of patients that receive moderately emetogenic chemotherapy, and
* (ii) patient preference for dexamethasone or placebo.

We will evaluate control of nausea and vomiting and the impact of both the side effects of dexamethasone and of nausea and vomiting on QOL. Therapy for acute emesis will be standardised (single dose intravenous granisetron and dexamethasone) and all patients will receive granisetron for delayed emetic control. Each patient will be randomly allocated to receive either dexamethasone or placebo after the first cycle of chemotherapy, and crossed over to the other arm for the second cycle. Patients will complete questionnaires that evaluate QOL, symptoms associated with dexamethasone, and nausea and vomiting at baseline and one week after their intravenous chemotherapy; they will also record symptoms in a daily diary.

The primary outcome measures are patient preference and overall QOL. The secondary objectives are: (1) to compare complete protection from delayed vomiting and severity of nausea between those receiving dexamethasone and those receiving placebo; (2) to compare differences in the impact of nausea and vomiting on QOL in those receiving dexamethasone and those receiving placebo, and (3) to compare differences in symptoms that have been associated with dexamethasone (insomnia, anxiety, agitation, mood, etc.) between patients receiving dexamethasone and those receiving placebo.

Significance: Our study will evaluate whether the benefits of dexamethasone for delayed emetic control outweigh potential side effects in patients receiving moderately emetogenic chemotherapy. It addresses a problem that is important to the majority of patients receiving anticancer chemotherapy. If overall QOL is improved on dexamethasone, then it should be prescribed routinely. If QOL is reduced on dexamethasone, and patients prefer the placebo, then its use as an antiemetic after moderately emetogenic chemotherapy should be limited to patients who initially have poor control of emesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer who will receive their first cycle of non-cisplatin moderately emetogenic chemotherapy. The following regimens can be administered:

  * 14-day regimens dose dense
  * 21-day regimens:

    * Adriamycin and Cyclophosphamide (AC) + a Taxane (T) Other regimens are eligible as long as no cisplatin or other highly emetogenic agent is part of the regimen, and a moderately emetogenic agent is included.
* Aged > 18 years
* Performance status of 0-2 on the European Cooperative Oncology Group (ECOG) performance scale
* Full recovery from any post operative sequelae
* Patients on opioids are eligible as long as their doses are stable (no change to dose in the previous week) and they have no nausea or vomiting in the 24 hours prior to the study
* Informed signed consent

Exclusion Criteria:

* Patient has previously received chemotherapy
* Patient has received or will receive radiation therapy to the abdomen or pelvis in the week prior to treatment
* Nausea or vomiting in the 24 hour period prior to commencing chemotherapy
* Use of antiemetics within 24 hours of the study period
* Patient has an active infection (e.g. pneumonia) or any uncontrolled disease (e.g. diabetes, gastrointestinal obstruction), which in the opinion of the investigator might confound the results of the study or pose unwarranted risk. Patients with controlled diabetes are eligible.
* Patient currently uses any illicit drugs, including marijuana, or has current evidence of alcohol abuse as determined by the investigator.
* Patient is mentally incapacitated or has a significant emotional or psychiatric disorder that in the opinion of the investigator precludes study entry.
* Patient has a history of hypersensitivity or contraindication to granisetron or dexamethasone.
* Patient is taking any systemic corticosteroid therapy at any dose. Topical or inhaled steroids are permitted.
* Use of benzodiazepines in the 48 hours prior to the study period with the exception of a single dose if used for sleeping.
* Abnormal laboratory values:

  * Absolute neutrophil count < 1.5 X 10^9/L
  * Platelet count < 100 X 10^9/L
  * Liver transaminases > 2.5 X upper limit of normal
  * Bilirubin > 1.5 X upper limit of normal
  * Creatinine > 1.5 X upper limit of normal
* Patients who will receive a different chemotherapy regimen in Cycle 2 than in Cycle 1. Changes in the dose of the same chemotherapy agents are permitted if required for toxicity.
* Refusal to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Patient preference for the dexamethasone or the placebo arm as assessed by asking the patient whether they preferred treatment period 1 or treatment period 2 | dexamethasone for one cycle of chemotherapy and placebo for one cycle
Difference in QOL as assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30 for chemotherapy cycles 1 and 2 | dexamethasone for one cycle and placebo for one cycle

SECONDARY OUTCOMES:
Differences in nausea and vomiting by treatment period and regimen | post period 2
Impact of nausea and vomiting on QOL by Functional Living Index-Emesis (FLIE) score by treatment period and regimen | post period 2
Symptoms and signs associated with dexamethasone use by treatment period and regimen: insomnia, indigestion/epigastric discomfort, hiccups, appetite, agitation, acne/facial rash, oral candida, depression, weight changes, blood pressure | post period 2
Strength of preference for treatment cycle including dexamethasone compared to treatment cycle including placebo (Much better, Little better, No difference) | post period 2
Proportion of patients having a clinically significant improvement in QOL (defined as an improvement in EORTC QLQ-C30 of 10 points or more) during each treatment cycle | post period 2

CONTACTS AND LOCATIONS:
Overall Officials: Ian Tannock, MD PhD, Principal Investigator — University Health Network University of Toronto
Locations (2):
- Canada (2):
  - Mount SinaiHospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario